CLINICAL TRIAL: NCT01805908
Title: Imaging With 111In-Pertuzumab to Predict Response to Trastuzumab in HER2 Positive Metastatic or Locally Advanced Breast Cancer
Brief Title: Imaging With 111 Indium (111In)-Pertuzumab (PmAb) to Predict Response to Trastuzumab (TmAb) in Human Epidermal Growth Factor-2 (HER2) Positive Metastatic Breast Cancer (MBC) or Locally Advanced Breast Cancer (LABC)
Acronym: PETRA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual is very poor
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCOG-2011-PETRA
Record Dates: First submitted 2013-02-12; First posted 2013-03-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: metastatic; breast cancer; herceptin; imaging; tumour response; adenocarcinoma; SPECT-CT; pertuzumab; trastuzumab; locally advanced
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 111In-Pertuzumab + SPECT-CT (Experimental): Radiopharmaceutical 111In-labeled Pertuzumab given intravenously prior to SPECT-CT imaging.
  Interventions: Other: 111In-Pertuzumab + SPECT-CT

INTERVENTIONS:
Other: 111In-Pertuzumab + SPECT-CT — 111In-PmAb will be provided ready for injection in a vial by Dr. Reilly's laboratory.

SUMMARY:
The general objective of the study is to improve the care of women with Human Epidermal Growth Factor Receptor-2 (HER2) positive metastatic or locally advanced breast cancer by using a radio-labelled biomarker with whole body Single Photon Emission Computed Tomography (SPECT) imaging to predict who will respond to treatment with Trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic, locally recurrent (local recurrence not amenable to surgical resection of curative intent), or locally advanced (T3 or T4, any N, M0) adenocarcinoma of the breast.
2. Tumour HER2 positive by immunohistochemistry for HER2 protein over-expression or by Fluorescence in situ Hybridization (FISH) for HER2 gene amplification, as defined by American Society of Clinical Oncology/College of American Pathologists guidelines
3. Initiating treatment with TmAb
4. Clinically measurable disease (by RECIST for patients with metastatic disease).

Exclusion Criteria:

1. Male gender.
2. Less than 18 years of age.
3. Life expectancy < 12 weeks.
4. Only site of metastases is liver.
5. Eastern Cooperative Oncology Group (ECOG) performance status of > 2.
6. Currently receiving PmAb or lapatinib for treatment of MBC.
7. Having received TmAb as adjuvant therapy within the previous 6 months.
8. Required to receive another radiopharmaceutical during the first week of the study.
9. Hypersensitivity to monoclonal antibodies.
10. Left Ventricular Ejection Fraction (LVEF) < 50% at baseline (within 42 days of study registration) as determined by either echocardiogram (ECHO) or Multi-Gated Acquisition (MUGA) scan.
11. Hematology and/or biochemistry parameters outside acceptable ranges:

    * absolute neutrophil count <1,500 cells/mm3,
    * platelet count <100,000 cells/mm3,
    * hemoglobin <9 g/dL,
    * total bilirubin > upper limit of normal (ULN) (unless subject has documented Gilbert's Syndrome),
    * aspartate aminotransferase (AST) [serum glutamic oxaloacetic transaminase(SGOT)] and alanine aminotransferase (ALT) [serum glutamic pyruvate transaminase(SGPT)] >2.5 × ULN,
    * serum creatinine >2.0 mg/dL or 177 μmol/L,
    * alanine aminotransferase (ALP) >2.5 x ULN.
12. Known pregnancy or lactating female (e.g. positive serum beta-human chorionic gonadotropin (B-hCG) pregnancy test).
13. For women of childbearing potential, failure to agree to use a highly effective form of contraception (patient and/or partner, e.g., surgical sterilization) or two effective forms of contraception (a reliable barrier method in conjunction with spermicidal jelly, birth control pills, or contraceptive hormone implants) and to continue its use for the duration of study treatment.
14. Any condition, which in the investigator's opinion would not make the patient a suitable candidate for inclusion in the trial.
15. Participation in another clinical trial.
16. Inability to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in tumour SUV (Standardized Uptake Value) from baseline to Day 8. | 8 days
  The imaging outcome for exploring the association between imaging and clinical outcome is the percent change in tumour SUV from baseline to Day 8 (Day 8 SUV - baseline SUV) /baseline SUV times 100%. The Positron Emission Tomography Evaluation Response Criteria In Solid Tumours (PERCIST) criterion will be used to measure SUV change.
Safety attributable to 111In-Pertuzumab injections | 3 months
  The safety, i.e. toxicities, attributable to 111In-Pertuzumab injections will be evaluated using the National Cancer Institute (NCI) Common Termination for Adverse Events Version 4.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) and tumour and normal tissue localization properties of 111In-PmAb will be measured. | 3 months
  The pharmacokinetics of 111In-PmAb and tumour and normal tissue localization properties of 111In-PmAb will be measured. Standard PK parameters (t1/2 alpha, t1/2β, V1, Vss and CL) will be calculated.
Optimal mass dose of 111In-PmAb | 3 months
  The dose of 111In-PmAb that is associated with the optimal SPECT-CT images will be established.
Change in tumour SUV from Baseline to Day 36 | 3 months
  The imaging outcome for exploring the association between imaging and clinical outcome is the percent change in tumour SUV from baseline to Day 36 (Day 36 SUV - baseline SUV) /baseline SUV times 100%. The Positron Emission Tomography Evaluation Response Criteria In Solid Tumours (PERCIST) criterion will be used to measure SUV change.
Clinical response (complete or partial) to treatment will be measured using Response Evaluation Criteria In Solid Tumours (RECIST) criteria. | 3 months
  Clinical response (complete or partial) to treatment will be measured using Response Evaluation Criteria In Solid Tumours (RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levine, Principal Investigator — Ontario Clinical Oncology Group, McMaster University; Raymond Reilly, Principal Investigator — University of Toronto; Kathleen Pritchard, Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Lam K, Chan C, Done SJ, Levine MN, Reilly RM. Preclinical pharmacokinetics, biodistribution, radiation dosimetry and acute toxicity studies required for regulatory approval of a Clinical Trial Application for a Phase I/II clinical trial of (111)In-BzDTPA-pertuzumab. Nucl Med Biol. 2015 Feb;42(2):78-84. doi: 10.1016/j.nucmedbio.2014.09.011. Epub 2014 Oct 14. PMID 25459109